CLINICAL TRIAL: NCT04925284
Title: A Dose-Escalation and Expansion Study of the Safety and Pharmacokinetics of XB002 as Single-Agent and Combination Therapy in Subjects With Inoperable Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of XB002 in Subjects With Solid Tumors (JEWEL-101)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XB002-101
Record Dates: First submitted 2021-05-27; First posted 2021-06-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Cervical Cancer; SCCHN; Pancreatic Cancer; Esophageal SCC; Metastatic Castration-resistant Prostate Cancer; Triple Negative Breast Cancer; Hormone Receptor-positive Breast Cancer; Epithelial Ovarian Cancer; Endometrial Cancer; Tissue Factor-Expressing Solid Tumors
Keywords: ADC; Antibody drug conjugate; Tissue Factor; Auristatin; Nivolumab; bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Pancreatic Neoplasms; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Neoplasms; Carcinoma, Ovarian Epithelial; Endometrial Neoplasms | interventions — Nivolumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Dose-escalation followed by cohort-expansion in tumor-specific expansion cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- XB002 Single-Agent Dose-Escalation Cohorts (Experimental): Subjects (Cohort A) will accrue in cohorts of 3-12 subjects in a modified i3+3 design.
  Interventions: Drug: XB002
- XB002 Single-Agent Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in subjects with non-small cell lung cancer [NSCLC] (Cohort B), epithelial ovarian cancer (Cohort D), cervical cancer (Cohort E), SCCHN (Cohort F), pancreatic cancer (Cohort G), Esophageal SCC (Cohort H), metastatic castration-resistant prostate cancer (Cohort I), triple-negative breast cancer (Cohort J), hormone-receptor positive breast cancer (Cohort K), endometrial cancer (Cohort L) and tumor agnostic tissue factor-expressing solid tumors (Cohort M).
  Interventions: Drug: XB002
- XB002 + Nivolumab Dose Escalation Cohorts (Experimental): Subjects (Cohort AN) will accrue in cohorts of 3-12 subjects in a modified i3+3 design.
  Interventions: Drug: XB002; Drug: Nivolumab
- XB002 + Nivolumab Dose Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in subjects with non-small cell lung cancer [NSCLC] (Cohort BN), SCCHN (Cohort FN).
  Interventions: Drug: XB002; Drug: Nivolumab
- Experimental: XB002 + Bevacizumab Dose Escalation Cohorts (Experimental): Subjects (Cohort AB) will accrue in cohorts of 3-12 subjects in a modified i3+3 design.
  Interventions: Drug: XB002; Drug: Bevacizumab

INTERVENTIONS:
Drug: XB002 — IV administration of XB002
Drug: Nivolumab — IV administration of Nivolumab
  Arms: XB002 + Nivolumab Dose Escalation Cohorts; XB002 + Nivolumab Dose Expansion Cohorts
Drug: Bevacizumab — IV administration of bevacizumab
  Arms: Experimental: XB002 + Bevacizumab Dose Escalation Cohorts

SUMMARY:
This is a Phase 1, open-label, multicenter, dose-escalation and expansion study evaluating the safety, tolerability, PK, pharmacodynamics, and clinical antitumor activity of XB002 administered IV q3w alone and in combination with nivolumab or bevacizumab to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically and radiologically confirmed solid tumor that is inoperable, locally advanced, metastatic, or recurrent.
* Dose-Escalation Stage Cohorts A, AB, and AN: The subject has received at least one systemic standard life-prolonging therapy unless it does not exist, or available therapies are intolerable or no longer effective.
* Cohort-Expansion Stage (Cohorts B - M, BN, FN and HN): The subject has received standard life-prolonging therapies unless they do not exist, or available therapies are intolerable or no longer effective.
* Cohort-Expansion Stage Cohort B and BN (Non-small Cell Lung Cancer): Subjects with Stage IV NSCLC who have documented radiographic disease progression during or following their last systemic anticancer therapy.
* Cohort-Expansion Stage Cohort D (Epithelial Ovarian Cancer): Subjects with high-grade serous ovarian cancer, including primary peritoneal cancer (PPC) and fallopian tube cancer (FTC) who have platinum-resistant disease following treatment with platinum-containing chemotherapy.
* Cohort-Expansion Stage Cohort E (Cervical Cancer): Subjects with persistent, recurrent, or metastatic carcinoma of the uterine cervix who have documented radiographic disease progression during or following their last systemic anticancer therapy.
* Cohorts F and FN (SCCHN): Subjects with head and neck cancer (squamous cell histology) who have documented radiographic disease progression during or following their last systemic anticancer therapy. Allowed primary tumor locations are oral cavity, oropharynx, hypopharynx, glottic larynx. Note: Excluded are subjects with primary tumor site of the nasopharynx.
* Cohort G (Pancreatic Cancer): Subjects with pancreatic cancer (adenocarcinoma histology) who have documented radiographic disease progression during or following their last systemic anticancer therapy.
* Cohort H (Esophageal SCC): Subjects with esophageal cancer (squamous cell histology) who have documented radiographic disease progression during or following their last systemic anticancer therapy. Note: subjects with esophageal adenocarcinoma and adenocarcinoma of gastroesophageal junction (GEJ) are excluded.
* Cohort I (mCRPC): Subjects with metastatic, castration resistant adenocarcinoma of the prostate. Note: Neuroendocrine differentiation and other histological features are permitted if adenocarcinoma is the primary histology.
* Cohort J (TNBC): Subjects with triple-negative (estrogen receptor negative [ER-]/progesterone receptor negative [PR-]/ human epidermal growth factor receptor 2 negative [HER-2-]) breast cancer who have documented radiographic disease progression during or following their last systemic anticancer therapy for inoperable locally advanced or metastatic disease.
* Cohort K (HR + BC): Subjects with breast cancer that is hormone receptor-positive (ER+ and/or PR+) and HER-2-) and who have documented radiographic disease progression during or following their last systemic anticancer therapy for inoperable locally advanced or metastatic disease.
* Cohort L (Endometrial Cancer): Subjects with locally advanced, recurrent or metastatic endometrial cancer who have documented radiographic disease progression during or following their last systemic anticancer therapy.
* Cohort M (Tumor-Agnostic Tissue Factor-Expressing Solid Tumors): Subjects with solid tumors other than those designated in Cohorts B-L and those which express tissue factor. Participation in this cohort will be at selected sites and countries based on site feasibility assessment.
* Expansion Cohorts: Subjects must have measurable disease per RECIST 1.1 as determined by the Investigator, except for subjects with prostate cancer without soft tissue disease and subjects with primary brain tumors.
* Tumor tissue material collected no more than 3 years prior to consent, if possible. If archival tumor tissue is not available, a fresh tumor biopsy may be collected from subjects enrolled in the Dose-Escalation Stage and should be collected from subjects in the Cohort-Expansion Stage.
* Recovery to baseline or ≤ Grade 1 severity (Common Terminology Criteria for Adverse Events version 5 [CTCAE v5]) from AEs.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ and marrow function.
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception.
* Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* Receipt of prior therapies as defined in study protocol
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
* Uncontrolled, significant intercurrent or recent illness.
* Major surgery within 4 weeks before first dose of study treatment
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG).
* Pregnant or lactating females
* Previously identified allergy or hypersensitivity to components of study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies.
* Another unresolved malignancy or a malignancy that is considered to be cured within 2 years before first dose of study treatment. Note: Subjects with superficial non-melanoma skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy within 2 years before first dose of study treatment are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Dose-Escalation Stage: MTD/recommended dose for XB002 | 18 months
  To determine the MTD and/or RD for further evaluation of IV administration of XB002 alone and in combination therapy in subjects with advanced malignancies
Cohort-Expansion Stage: Objective Response Rate (ORR) | 12 months
  To evaluate preliminary efficacy of XB002 when administered alone and in combination therapy by determining the ORR per RECIST 1.1 (or other applicable response criteria eg. RANO or PCWG3 criteria) as assessed by the Investigator

SECONDARY OUTCOMES:
Safety of XB002: Adverse Events | 30 months
  To evaluate the safety of XB002 through the evaluation of incidence and severity of nonserious adverse events (AEs) and serious adverse events (SAEs)
Tolerability of XB002 as evaluated by the duration of exposure for the study | 30 months
  To evaluate the tolerability of XB002 through the evaluation of duration of exposure for the study treatment
Tolerability of XB002 as evaluated dose intensity of the study treatment | 30 months
  To evaluate the tolerability of XB002 through the evaluation of dose intensity of the study treatment
Maximum Plasma Concentration (Cmax) | 30 months
  To evaluate the Cmax for XB002, total antibody, and free payload at scheduled visits over time
Trough Concentration (Ctrough) | 30 months
  To evaluate the Ctrough of XB002, total antibody, and free payload at scheduled visits over time
Immunogenicity of XB002 | 30 months
  To assess the immunogenicity of XB002 as measured by anti-drug antibody (ADA) analysis
Anti-tumor activity of XB002: Objective Response Rate (ORR) | 30 months
  To evaluate the anti-tumor activity of XB002, as measured by ORR, per RECIST 1.1 (or other applicable response criteria eg. RANO or PCWG3 criteria) as assessed by the Investigator (dose escalation stage) or by a BIRC for selected cohorts (cohort expansion stage).
Anti-tumor activity of XB002: Duration of Response (DOR) | 30 months
  To evaluate the anti-tumor activity of XB002, as measured by DOR, per RECIST 1.1 (or other applicable response criteria eg. RANO or PCWG3 criteria) as assessed by the Investigator (dose escalation stage) or by a BIRC for selected cohorts (cohort expansion stage)
Anti-tumor activity of XB002: Progression Free Survival (PFS) | 30 months
  To evaluate the anti-tumor activity of XB002, as measured by PFS, per RECIST 1.1 (or other applicable response criteria eg. RANO or PCWG3 criteria) as assessed by the Investigator (dose escalation stage) or by a BIRC for selected cohorts (cohort expansion stage)
Cohort-Expansion Stage: overall survival | 12 months
  To evaluate overall survival

CONTACTS AND LOCATIONS:
Locations (95):
- United States (34):
  - Exelixis Clinical Site #48, Birmingham, Alabama
  - Exelixis Clinical Site #20, Tucson, Arizona
  - Exelixis Clinical Site#95, Tucson, Arizona
  - Exelixis Clinical Site#58, Little Rock, Arkansas
  - Exelixis Clinical Site#59, Fountain Valley, California
  - Exelixis Clinical Site #21, Los Angeles, California
  - Exelixis Clinical Site #26, Los Angeles, California
  - Exelixis Clinical Site #16, New Haven, Connecticut
  - Exelixis Clinical Site #22, Washington D.C., District of Columbia
  - Exelixis Clinical Site#93, Chicago, Illinois
  - Exelixis Clinical Site #6, Baltimore, Maryland
  - Exelixis Clinical Site #18, Columbia, Maryland
  - Exelixis Clinical Site #25, Boston, Massachusetts
  - Exelixis Clinical Site #19, Detroit, Michigan
  - Exelixis Clinical Site #10, Detroit, Michigan
  - Exelixis Clinical Site #5, St Louis, Missouri
  - Exelixis Clinical Site #11, Omaha, Nebraska
  - Exelixis Clinical Site #8, East Brunswick, New Jersey
  - Exelixis Clinical Site #7, New Brunswick, New Jersey
  - Exelixis Clinical Site #23, Albany, New York
  - Exelixis Clinical Site#67, Lake Success, New York
  - Exelixis Clinical Site #12, New York, New York
  - Exelixis Clinical Site #15, Cleveland, Ohio
  - Exelixis Clinical Site #29, Cleveland, Ohio
  - Exelixis Clinical Site #49, Hilliard, Ohio
  - Exelixis Clinical Site #4, Oklahoma City, Oklahoma
  - Exelixis Clinical Site #3, Nashville, Tennessee
  - Exelixis Clinical Site #24, Austin, Texas
  - Exelixis Clinical Site #1, Austin, Texas
  - Exelixis Clinical Site #32, Dallas, Texas
  - Exelixis Clinical Site #14, Dallas, Texas
  - Exelixis Clinical Site#92, Houston, Texas
  - Exelixis Clinical Site #2, San Antonio, Texas
  - Exelixis Clinical Site #9, Charlottesville, Virginia
- Australia (5):
  - Exelixis Clinical Site#75, Miranda, New South Wales
  - Exelixis Clinical Site#70, Nedlands, Western Australia
  - Exelixis Clinical Site #37, Darlinghurst
  - Exelixis Clinical Site #44, Liverpool
  - Exelixis Clinical Site #35, Saint Leonards
- Belgium (6):
  - Exelixis Clinical Site#71, Charleroi, Hainaut
  - Exelixis Clinical Site#66, Liège, Liege
  - Exelixis Clinical Site#56, Brussels
  - Exelixis Clinical Site #30, Brussels
  - Exelixis Clinical Site #47, Edegem
  - Exelixis Clinical Site #38, Ghent
- France (8):
  - Exelixis Clinical Site#69, Lyon, Auvergne-Rhône-Alpes
  - Exelixis Clinical Site #45, Bordeaux
  - Exelixis Clinical Site #41, Pierre-Bénite
  - Exelixis Clinical Site#68, Poitiers
  - Exelixis Clinical Site #50, Rennes
  - Exelixis Clinical Site#63, Strasbourg
  - Exelixis Clinical Site#53, Villejuif
  - Exelixis Clinical Site#87, Paris, Île-de-France Region
- Italy (8):
  - Exelixis Clinical Site#62, Milan, MI
  - Exelixis Clinical Site #54, Ancona
  - Exelixis Clinical Site#60, Florence
  - Exelixis Clinical Site#84, Milan
  - Exelixis Clinical Site #40, Roma
  - Exelixis Clinical Site#90, Roma
  - Exelixis Clinical Site #34, Rozzano
  - Exelixis Clinical Site#61, Siena
- Netherlands (4):
  - Exelixis Clinical Site#73, Amsterdam, North Holland
  - Exelixis Clinical Site#76, Rotterdam, South Holland
  - Exelixis Clinical Site#65, Groningen
  - Exelixis Clinical Site #39, Maastricht
- South Korea (10):
  - Exelixis Clinical Site#79, Anyang-si, Gyeonggi-do
  - Exelixis Clinical Site#80, Seongnam-si, Gyeonggi-do
  - Exelixis Clinical Site#74, Seongnam-si, Gyeonggido
  - Exelixis Clinical Site#83, Suwon, Gyeonggido
  - Exelixis Clinical Site#86, Pusan, Gyeongsangnam-do
  - Exelixis Clinical Site#78, Hwasun, Jeonranamdo
  - Exelixis Clinical Site#77, Seoul, Seoul Teugbyeolsi
  - Exelixis Clinical Site#94, Seoul, Seoul Teugbyeolsi
  - Exelixis Clinical Site#81, Seoul, Seoul Teugbyeolsi
  - Exelixis Clinical Site#85, Seoul, Seoul Teugbyeolsi
- Spain (14):
  - Exelixis Clinical Site #27, Barcelona
  - Exelixis Clinical Site #36, Barcelona
  - Exelixis Clinical Site#55, Barcelona
  - Exelixis Clinical Site#82, Barcelona
  - Exelixis Clinical Site #31, Lleida
  - Exelixis Clinical Site#64, Madrid
  - Exelixis Clinical Site #17, Madrid
  - Exelixis Clinical Site #33, Madrid
  - Exelixis Clinical Site #42, Madrid
  - Exelixis Clinical Site #13, Madrid
  - Exelixis Clinical Site #46, Málaga
  - Exelixis Clinical Site #43, Valencia
  - Exelixis Clinical Site #51, Valencia
  - Exelixis Clinical Site#72, Zaragoza
- United Kingdom (6):
  - Exelixis Clinical Site#88, Leicester, England
  - Exelixis Clinical Site#89, London, England
  - Exelixis Clinical Site#91, Cardiff, Wales
  - Exelixis Clinical Site #52, Glasgow
  - Exelixis Clinical Site#57, London
  - Exelixis Clinical Site #28, Newcastle upon Tyne